CLINICAL TRIAL: NCT00431002
Title: Provincial Roll-Out Bone Health Strategy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Maureen C. Ashe, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H05-70624
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Osteoporosis
Keywords: Exercise; Resistance training
MeSH Terms: conditions — Osteoporosis; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Resistance training — See Detailed Description.

SUMMARY:
The main purpose of this study is to investigate the effect of two different group-based exercise programs on fall risk (muscular strength and balance) and bone strength in older women aged over 65-75 years who have low bone mass. We are also trying to determine if once a week exercise is as effective on health outcomes as twice a week. We hypothesize that twice a week exercise will be more effective than once a week or sham exercise.

ELIGIBILITY:
Inclusion Criteria:

* inactive (less than twice weekly exercising) women aged 65-75 years old

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2008-09

PRIMARY OUTCOMES:
Physiologic Profile Assessment (Fall Risk)

SECONDARY OUTCOMES:
Bone strength using peripheral quantitative computed tomography (pQCT)

CONTACTS AND LOCATIONS:
Overall Officials: K M Khan, PhD, Principal Investigator — University of British Columbia